CLINICAL TRIAL: NCT03093272
Title: A Phase 2 Study of Docetaxel Plus Apalutamide in Castration-Resistant Prostate Cancer Patients Post Abiraterone Acetate
Brief Title: A Study of Docetaxel + ARN-509 in Castration-Resistant Prostate Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Safety concerns
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Janssen Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Lauren C. Harshman, Assistant Professor of Medicine, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16-485
Record Dates: First submitted 2017-03-15; First posted 2017-03-28 (Actual); Results first posted 2020-03-30 (Actual); Last update posted 2020-04-09 (Actual); Status verified 2020-04

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Leuprolide; Prednisone; Docetaxel; apalutamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ARN-509 Combined With Docetaxel (Experimental): * Apalutamide (ARN-509) will be taken orally at home daily
  * Docetaxel will be administered every 3 weeks intravenously
  * Prednisone will be taken orally twice daily
  * Leuprolide Acetate will be administered at the specification of the physician
  Interventions: Drug: Leuprolide Acetate; Drug: Prednisone; Drug: Docetaxel; Drug: Apalutamide

INTERVENTIONS:
Drug: Leuprolide Acetate — a GnRH agonist
  Other Names: Lupron Injection
Drug: Prednisone — Prednisone is a corticosteroid
  Other Names: Deltasone
Drug: Docetaxel — Docetaxel is an antineoplastic agent that acts by disrupting the microtubular network in cells that is essential for mitotic and interphase cellular functions. Docetaxel binds to free tubulin and promotes the assembly of tubulin into stable microtubules while simultaneously inhibiting their disassembly.
  Other Names: Docefrez; Taxotere
Drug: Apalutamide — The apalutamide drug substance is an almost white to slightly brown powder. The tablet formulation of apalutamide is an immediate release oral tablet containing 60-mg of drug substance, with a non-functional green film coat
  Other Names: ARN-509

SUMMARY:
This research study is studying a combination of drugs as a possible treatment for castration-resistant prostate cancer.

The interventions involved in this study are:

* Docetaxel (a type of chemotherapy)
* Apalutamide (the study medication, also known as ARN-509)
* Prednisone (a corticosteroid given to prevent reactions to docetaxel).
* Leuprolide acetate (also known as Lupron, a GnRH agonist or similar drug which is standard of care, causes chemical castration which greatly lowers the level of testosterone in the body)

DETAILED DESCRIPTION:
This research study is a Phase II clinical trial. Phase II clinical trials test the safety and effectiveness of an investigational intervention to learn whether the intervention works in treating a specific disease. "Investigational" means that the intervention is being studied.

Apalutamide is considered an investigational product, which is believed to reduce the growth of prostate cancer cells. The FDA (the U.S. Food and Drug Administration) has not approved apalutamide as a treatment for any disease, but it is being studied in prostate cancer. Docetaxel is an approved therapy for this type of cancer. The FDA has not approved the combination of the two drugs in any use.

In this research study, the investigators are evaluating the combination of two drugs, docetaxel with apalutamide. The investigators will keep track of participants' prostate-specific antigen (PSA), scans, and overall health to determine how well this drug combination works at treating this type of cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed adenocarcinoma of the prostate
* Castration-resistant prostate cancer requires the following criteria:

  * A castrate level of testosterone (< 50ng/dL)
  * Prostate cancer progression on or since last treatment as documented by PSA rise or bone progression according to PCWG2 or soft tissue radiographic progression according to RECIST criteria Version 1.1
  * If on anti-androgen, will need to show no PSA decline after at least a 6 week withdrawal period from the last dose of bicalutamide or nilutamide or 4 weeks from last flutamide dose
  * Will require a 2 week washout period from last dose of ketoconazole, abiraterone acetate or radiation
* Treatment with abiraterone acetate for CRPC in the past is required. Does not need to be the last treatment prior to enrollment.
* There is no limit to number of prior therapies
* Metastatic disease by bone scan or other nodal or visceral lesions on CT or MRI
* Age ≥ 18 years
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 (See Appendix A)
* Adequate organ function as evaluated by the following laboratory criteria:

  * Hemoglobin ≥ 9g/dL; no transfusions and erythropoietin supplementation permitted within the last 3 months
  * Absolute neutrophil count (ANC) ≥ 1500/µL
  * Platelet count ≥ 100 x 10^9/L
  * Total bilirubin ≤ upper limit of normal (ULN, Note: In subjects with Gilbert's syndrome, if total bilirubin is ≥ 1.5 × ULN, measure direct and indirect bilirubin and if direct bilirubin is ≤ ULN, subject may be eligible)
  * AST and ALT < 2.5 x ULN or < 5x the ULN if liver metastasis
  * Serum creatinine < 2.0 × ULN or creatinine clearance > 30cc/min
  * Serum albumin ≥ 3.0 g/dL
  * Serum potassium ≥ 3.5 mmol/L (if < 3.5, can be repleted and reassess for eligibility as long as stable off potassium supplementation for > 48 hrs)
* Ability to swallow the study drug as a whole tablet
* The effects of apalutamide and docetaxel on the developing human fetus are unknown. For this reason and because chemotherapeutic agents are known to be teratogenic, men must agree to use adequate contraception. Specifically, they must agree to use a condom (even men with vasectomies) and another effective method of birth control if he is having sex with a woman of childbearing potential or agree to use a condom if he is having sex with a woman who is pregnant while on study drug and for 3 months following the last dose of study drug. They must also agree not to donate sperm during the study and for 3 months after receiving the last dose of study drug.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Pathology consistent with majority of specimen having small cell carcinoma of the prostate (prostate cancer with neuroendocrine features is acceptable).
* Prior treatment with enzalutamide for CPRC; non-CRPC use allowed (e.g., neoadjuvant, combined with radiation for localized disease and didn't progress while on it in those settings)
* Prior treatment with docetaxel chemotherapy except if > 12 months since it was given in either the neoadjuvant or adjuvant setting or for hormone sensitive disease (e.g., CHAARTED population)
* Presence of untreated brain metastasis
* Seizure or known condition that may pre-dispose to seizure (including but not limited to prior stroke, transient ischemic attack within 1 year prior to randomization, brain arteriovenous malformation; or intracranial masses such as schwannomas and meningiomas that are causing edema or mass effect). Loss of consciousness within 12 months may be permitted upon discussion with study PI.
* Medications known to lower the seizure threshold must be discontinued or substituted at least 4 weeks prior to study entry.
* Current, recent (within 4 weeks of the first dose of this study), or planned participation in an experimental drug study
* Persistent grade > 1 (NCI CTCAE v4.0) AEs due to investigational drugs that were administered more than 14 days before study enrollment.
* Radiation within 2 weeks prior to entering the study
* Peripheral neuropathy ≥ Grade 2.
* Current evidence of any of the following:

  * Uncontrolled hypertension
  * Gastrointestinal disorder affecting absorption
  * Active infection (e.g., human immunodeficiency virus [HIV] or viral hepatitis) or other medical condition that would make prednisone/prednisolone (corticosteroid) use contraindicated
* Uncontrolled intercurrent illness including, but not limited to, severe or unstable angina, myocardial infarction, symptomatic congestive heart failure (defined as New York Heart Association Grade II or greater), arterial or venous thromboembolic events (e.g., pulmonary embolism), or clinically significant ventricular arrhythmias, significant vascular disease (e.g. aortic aneurysm, aortic dissection), or symptomatic peripheral vascular disease within 6 months prior to randomization.
* Psychiatric illness/social situations that would limit compliance with study requirements.
* Any condition that in the opinion of the investigator, would preclude participation in this study
* History of allergic reactions or severe hypersensitivity reactions to drugs formulated with polysorbate 80 or antisense oligonucleotides.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to apalutamide or docetaxel
* Participants receiving any medications or substances that are strong inhibitors or inducers of CYP3A4 are ineligible. Because the lists of these agents are constantly changing, it is important to regularly consult a frequently-updated list such as http://medicine.iupui.edu/clinpharm/ddis/table.aspx; medical reference texts such as the Physicians' Desk Reference may also provide this information. As part of the enrollment/informed consent procedures, the patient will be counseled on the risk of interactions with other agents, and what to do if new medications need to be prescribed or if the patient is considering a new over-the-counter medicine or herbal product.
* Inability to comply with study and/or follow-up procedures

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2017-06-23 (Actual); Primary Completion 2019-05-16 (Actual); Study Completion 2019-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lauren C Harshman, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Apalutamide Combined With Docetaxel: * Apalutamide (ARN-509): 240mg (four 60mg tablets), oral, once daily
  * Docetaxel: 75mg/m2 in 250cc Normal Saline, IV, every 21 days (3 weeks)
  * Prednisone: 5mg, oral, twice daily
Period: Overall Study
Arm/Group | Apalutamide Combined With Docetaxel
Started | 9
Completed | 9
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Apalutamide Combined With Docetaxel
Number analyzed (Participants) | 9
Age, Customized [Count of Participants; unit: Participants]
  <60 | 1
  60-69 | 3
  70-79 | 4
  80-89 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 9
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: White | 8
  Race/Ethnicity: Hispanic | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 9
Prior treatment with abiraterone acetate [Count of Participants; unit: Participants] | 9
Duration on abiraterone acetate [Median (Full Range); unit: months] | 5.5 [2.4 to 37.1]
Time interval between abiraterone acetate initiation and protocol treatment [Median (Full Range); unit: months] | 6.0 [2.9 to 37.9]
ECOG performance status [Count of Participants; unit: Participants] — The ECOG Scale of Performance Status is a standard criteria scale for measuring how the disease impacts a patient's daily living abilities. It describes a patient's level of functioning in terms of their ability to care for themself, daily activity, and physical ability (walking, working, etc.). The scale ranges from 0 to 5, with 0 being fully active and able to carry on all pre-disease performance without restriction and 5 being dead.
  Participants
    Performance Status 0 | 7
    Performance Status 1 | 2
Gleason score [Count of Participants; unit: Participants] — The Gleason Score is the grading system used to determine the aggressiveness of prostate cancer based on pathological review. Typical Gleason Scores range from 6-10. The higher the Gleason Score, the more aggressive the cancer.
  Participants
    Gleason Score 6 | 1
    Gleason Score 7 | 0
    Gleason Score 8-10 | 7
    Gleason Score Missing | 1
PSA level [Median (Full Range); unit: ng/mL] | 48.3 [0.4 to 969.8]
Number of Patients with Disease in Specific Sites [Count of Participants; unit: Participants] — It is summarized regardless of target or non-target lesions. Patients may have more than 1 site, therefore, the percentage was calculated based on 9.
  Participants
    Bone | 8
    Lymph Nodes | 6
    Prostate | 1
    Liver | 1
    Others | 2

OUTCOME MEASURES:

1. Primary Outcome: To Evaluate Progression-free Survival on the Combination of Docetaxel Plus Apalutamide
Description: Progression free survival (PFS) is defined as the time from treatment initiation until the occurrence of one of the following:
  1. A participant was considered to have progressed by bone scan if
     1. the first bone scan with greater than or equal to (≥) 2 new lesions compared to baseline was observed in less than (<) 12 weeks from study drug initiation and was confirmed by a second bone scan taken ≥6 weeks later showing ≥2 additional new lesions (a total of ≥4 new lesions compared to baseline);
     2. the first bone scan with ≥2 new lesions compared to baseline was observed in ≥12 weeks from study drug initiation and the new lesions were verified on the next bone scan ≥6 weeks later (a total of ≥2 new lesions compared to baseline);
  2. Progression of soft tissue lesions measured by computerized tomography (CT) or magnetic resonance imaging (MRI) by RECIST v. 1.1; or
  3. Death from any cause.
Time Frame: Disease was evaluated radiologically at baseline and every 12 weeks on treatment; PFS follow up was up to 9.4 months
Population: Three patients did not have the progression defined by protocol (patients 1, 2, and 8). Two patients (patients 2 and 8) did not have follow-up scans, and thus PFS was censored at the date of the registration. One patient (patient 1) progressed via rising PSA, not radiographically.
Measure: Number; unit: months
Arm/Group | Apalutamide Combined With Docetaxel
Number analyzed (Participants) | 9
months
  Participant 1 | 5.6
  Participant 2 | NA — Patient did not have follow up scans to document PFS.
  Participant 3 | 5.6
  Participant 4 | 8.1
  Participant 5 | 1.8
  Participant 6 | 4.8
  Participant 7 | 5.1
  Participant 8 | NA — Patient did not have follow up scans to document PFS.
  Participant 9 | 9.4

2. Secondary Outcome: Number of Participants With Dose-Limiting Toxicities in the Safety Lead-in Group (First 6 Patients)
Description: Specific adverse events will be recorded during the safety lead-in phase of 6 patients. Any toxicities considered unacceptable during this time will be considered a dose-limiting toxicity and will be summarized among all patients evaluable for a dose-limiting toxicity (DLT).
Time Frame: First 3 weeks of treatment
Population: If the first 3 patients were accrued had no DLTs, then an additional 3 patients were accrued to observe for DLTs. If less than 2 patients experienced a DLT, the study opened to full accrual.
Measure: Count of Participants; unit: Participants
Arm/Group | Apalutamide Combined With Docetaxel
Number analyzed (Participants) | 6
Participants
  Dose-limiting toxicity identified | 0
  No dose-limiting toxicity identified | 6

3. Secondary Outcome: Maximum Blood Concentration (Cmax) for Docetaxel Pharmacokinetic Analysis
Description: The pharmacokinetic (PK) parameters of the first 9 patients enrolled at Dana-Farber Cancer Institute will be determined using noncompartmental methods with WinNonLin version 5.2. Maximum blood concentration (Cmax) will be determined by visual inspection. Due to the premature termination of the study, only 9 patients were evaluated. The PK samples were collected on Days 1 and 2 of the first two treatment cycles.
Time Frame: Cycle 1, 2: During infusion at pre-dose, 15 minutes and 30 minutes post-dose, end of dose, and 0.5, 1, 1.5, 2, 4, 6, 8, 24 hours post dose.
Population: Pharmacokinetic samples were not collected or received for 3 patients during C2D1.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Apalutamide Combined With Docetaxel
Number analyzed (Participants) | 9
ng/mL
  Cycle 1 | 2415 (970)
  Cycle 2: number analyzed (Participants) | 6
  Cycle 2 | 1641 (867)

4. Secondary Outcome: Area Under the Curve (AUC) for Docetaxel Pharmacokinetic Analysis
Description: The area under the blood concentration-time curve (linear trapezoidal rule) will be determined between 0-24 hours (AUC0-24). The PK samples were collected during the first two days of cycles 1 and 2.
Time Frame: as for outcome 3
Population: Pharmacokinetic samples were not collected or received for 3 patients during C2D1.
Measure: Mean (Standard Deviation); unit: ng•h/mL
Arm/Group | Apalutamide Combined With Docetaxel
Number analyzed (Participants) | 9
ng•h/mL
  Cycle 1 | 3406 (1426)
  Cycle 2: number analyzed (Participants) | 6
  Cycle 2 | 3095 (1407)

5. Secondary Outcome: Serum PSA Change From Baseline to 12 Weeks on Treatment
Description: The maximum percent PSA change (rise or fall) from baseline to after 12 weeks on study. For patients who discontinue on or before the 12 week assessment or for whom the 12 week assessment is missing, the last observation prior to the week 12 assessment will be utilized. Patients with no post-baseline PSA data will be excluded from the summary.
Time Frame: PSA was measured on Cycle 1 Day 1 (Baseline) and at 12 weeks on treatment.
Measure: Median (Inter-Quartile Range); unit: percent
Arm/Group | Apalutamide Combined With Docetaxel
Number analyzed (Participants) | 9
percent | 13.0 [-36.3 to 28.8]

6. Secondary Outcome: Overall Survival
Description: Overall Survival (OS) is defined as the time from trial treatment start to death due to any cause, or censored at date last known alive.
Time Frame: Measured from end of study treatment to death due to any cause; OS measured as 22.4 months
Measure: Number; unit: months
Arm/Group | Apalutamide Combined With Docetaxel
Number analyzed (Participants) | 9
months
  Participant 1 | 22.4
  Participant 2 | 4.2
  Participant 3 | 21.2
  Participant 4 | 16.8
  Participant 5 | 1.8
  Participant 6 | 9.0
  Participant 7 | 10.1
  Participant 8 | 5.9
  Participant 9 | 12.2

ADVERSE EVENTS:
Time Frame: Participants were assessed for adverse events on days 1, 8 and 15 for cycle 1, on days 1 and 15 for cycle 2, and every cycle thereafter; Treatment duration was up to 12 cycles in this study (1 cycle=21 days).
Description: Maximum grade toxicity by type was first calculated. Serious adverse events were defined as any untoward medical occurrence based on ICH and EU Guidelines on Pharmacovigilance for Medicinal Products for Human Use
Arm/Group | Apalutamide Combined With Docetaxel
All-Cause Mortality (participants affected / at risk) | 1/9
Serious Adverse Events (participants affected / at risk) | 4/9
Other Adverse Events (participants affected / at risk) | 9/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Apalutamide Combined With Docetaxel (N=9)
Infusion related reaction (General disorders) | 1
Neutrophil count decreased (Investigations) | 2
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Apalutamide Combined With Docetaxel (N=9)
Hyperthyroidism (Endocrine disorders) | 1
Hypothyroidism (Endocrine disorders) | 1
Eye disorders - Other, specify - Blepharitis (Eye disorders) | 1
Diarrhea (Gastrointestinal disorders) | 2
Enterocolitis (Gastrointestinal disorders) | 1
Mucositis oral (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 3
Vomiting (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 4
Fever (General disorders) | 1
General disorders and administration site conditions - Other, specify - Infusion Related Reaction (General disorders) | 1
General disorders and administration site conditions - Other, specify - Rhinorrhea (General disorders) | 1
Infusion related reaction (General disorders) | 3
Paronychia (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Alkaline phosphatase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 1
Neutrophil count decreased (Investigations) | 4
Urine output decreased (Investigations) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Dysgeusia (Nervous system disorders) | 2
Peripheral sensory neuropathy (Nervous system disorders) | 2
Insomnia (Psychiatric disorders) | 2
Urinary incontinence (Renal and urinary disorders) | 1
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 3
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1
Rash acneiform (Skin and subcutaneous tissue disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1
Skin/subcutaneous tissue disorders; Other, specify - Nail Changes (Skin and subcutaneous tissue disorders) | 1
Skin/subcutaneous tissue disorders; Other, specify - Rash (Skin and subcutaneous tissue disorders) | 1
Skin/subcutaneous tissue disorders; Other, specify - Rash - Unspecified (Skin and subcutaneous tissue disorders) | 1
Skin/subcutaneous tissue disorders; Other, specify - Tearing (Skin and subcutaneous tissue disorders) | 1
Hypertension (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-06-15): https://cdn.clinicaltrials.gov/large-docs/72/NCT03093272/Prot_SAP_000.pdf